CLINICAL TRIAL: NCT03628222
Title: Transbronchial Lung Biopsy Guided by Electromagnetic Navigation Bronchoscopy: A Prospective, Randomized, Multicenter, Superiority Study
Brief Title: Transbronchial Lung Biopsy Guided by ENB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changzhou LungHealth Medtech Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LHCTP001
Record Dates: First submitted 2018-07-23; First posted 2018-08-14 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lung Lesion(s) Requiring Evaluation
Keywords: Lung lesion; Electromagnetic navigation bronchoscopy (ENB); Transbronchial lung biopsy(TBLB); bronchoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENB-TBLB (Experimental): Under ENB guidance, the Location Catheter and Guide Catheter reach the lesion. After confirmation by X-ray, biopsy tools are introduced and specimens are obtained.
  Interventions: Device: ENB-TBLB
- X-ray-TBLB (Active Comparator): Based on chest CT, the physician determines the lesion location. Under X-ray guidance, via the bronchoscope's working channel, the biopsy forceps and brush are introduced and specimens are obtained.
  Interventions: Device: X-ray-TBLB

INTERVENTIONS:
Device: ENB-TBLB — ENB Guidance: The iLungTM SuperNavigator system will be used, it comprises of iLungTM ENB system, location catheter and guide catheter. The guide catheter can supply a 1.9 mm working channel for biopsy tools.
  The location catheter is inserted into the guide catheter beforehand, then both are introduced via the working channel of the bronchoscope. Under guidance of ENB system, the location catheter reaches the lesion, and actual distance is confirmed by the X-ray.
  TBLB: Location catheter is retracted, then the biopsy forceps and brush was introduced, and pathologic specimens are obtained.
  Arms: ENB-TBLB
Device: X-ray-TBLB — Based on chest CT, the physician determines the lesion location. Under X-ray guidance, via the bronchoscope's working channel, the biopsy forceps and brush are introduced and pathologic specimens are obtained.
  Arms: X-ray-TBLB

SUMMARY:
The purpose of this study is to evaluate the performance and safety of electromagnetic navigation bronchoscopy (ENB) system and system kit (iLungTM SuperNavigator) .

DETAILED DESCRIPTION:
This is prospective, randomized, multicenter, superiority study. 8 top centers in China was chosen. Subject which has peripheral lung lesions (PLLs) detected by chest CT scan, requires biopsy diagnosis, and meets all inclusion and exclusion criteria, will be included in this trial. Firstly physician determines the lesion biopsied, then the subject will be randomized to experimental or control group. The experimental group is treated with ENB guided transbronchial lung biopsy (TBLB)(ENB-TBLB): Under ENB guidance, the location sensor reaches the edge of the lesion, and X-ray is used for actual distance confirmation, if physician determines the distance is enough for biopsy, TBLB will be conducted. The control group will be treated with TBLB using X-ray guidance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older;
* Subject presents with PLL(s) detected by chest CT scan and biopsy diagnosis is needed;
* Subject is willing to receive bronchoscopy voluntarily, and meets relevant requirements;
* Subject or their guardian understands the purpose of this trial, and willing to participate in the trial voluntarily and sign Informed Consent Form (ICF).

Exclusion Criteria:

* Subject has participated in a drug or device study (drug study within 3 months or device study within 1 month);
* Female subject who is pregnant or nursing;
* Allergic to anesthetic;
* Bronchoscopy contraindications, include: Active hemoptysis; Newly developed myocardial infarction or unstable angina attack; Severe cardiac and pulmonary dysfunction; Severe hypertension and arrhythmia; Uncorrectable bleeding tendency (Such as severe clotting dysfunction, uremia, and severe pulmonary hypertension, etc.); Severe superior vena cava obstructive syndrome; Suspected aortic aneurysm; Multiple lung bullae; Extremely exhausted systemic conditions;
* Subject with serious lung disease (Such as: severe bronchiectasis, severe emphysema, etc) ,which investigator considers not appropriate for this examination;
* Subject with implanted pacemaker or defibrillator;
* Lack of patient cooperation for bronchoscopy, such as patient with mental disorders, dysgnosia, psychological disorder etc;
* Conditions investigator considers not appropriate for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Compare the diagnostic yield of ENB-TBLB with that of X-ray-TBLB | Up to 6 months
  Diagnostic yield = Lesions with definitive diagnosis /total lesions with biopsies.
  Comment: Lesions with definitive diagnosis: 1. Biopsy pathologic results show as benign or malignant lesion (fungi, tuberculosis, or nodule disease,etc.); 2. Biopsy pathologic results are abnormal lung tissue, but through later diagnosis, treatment and other observation measures, the lesion is proved to be benign; 3. When the patient cannot be diagnosed after a 6-month following-up, a CT or enhanced CT scan is needed and the physician make a final diagnosis based on the scan results.

SECONDARY OUTCOMES:
Incidence of navigation success | At 1 day of ENB procedure
  This outcome just apply to experimental group. Incidence of navigation success = the number of lesions navigated successfully/total lesions with ENB procedure × 100%.
  Criteria for navigation success: When the navigation software shows the distance of location sensor to the target ≤10mm, using X-ray to confirm the actual distance, if the physician determine that biopsy can be conducted, the navigation is successful, if not, the navigation fails.
Lesion detection rate | About 3-7days after ENB or X-ray procedure
  Based on the biopsy pathologic results, evaluate the lesion detection rate of experimental and control group.
  Lesion detection rate = Total lesions detected / Total lesions with biopsies. Comment: 'Lesions detected' indicates pathologic result shows as abnormal lung tissue.
Navigation time | At 1 day of ENB or X-ray procedure
  Evaluate navigation time of experimental and control group. Experimental group: After registration, the location sensor returns the carina. Navigation begins from the carina and ends when the sensor reaches the edge of the lesion, which is verified by the X-ray. This period is defined as navigation time of experimental group.
  Control group: Under X-ray guidance, the bronchoscope moves from the carina to the edge of the lesion. This period is defined as navigation time of control group.
Evaluate the user satisfaction of ENB system and system kit | At 1 day of ENB procedure
  After each ENB procedure, the investigator evaluate the operational performance of ENB system and system kit through a pre-designed questionnaire which includes terms related to the device function, convenience, reliability and safety.
The adverse events and device defects related to the ENB system and system kit | Up to 3 days
  Adverse events: Include incidence of pneumothorax, bleeding, respiratory failure, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Principal Investigator — The First Affiliate Hospital of Guangzhou Medical University
Locations (8):
- China (8):
  - Cancer Hospital, Chinese Academy of Medical sciences, Beijing, Beijing Municipality
  - The second affiliated hospital, Fujian Medical University, Quanzhou, Fujian
  - The First Affiliate Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The first affiliated hospital of Suzhou University, Suzhou, Jiangsu
  - Shanghai Chest hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - The first affiliated hospital, Zhejiang university, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahajan AK, Patel S, Hogarth DK, Wightman R. Electromagnetic navigational bronchoscopy: an effective and safe approach to diagnose peripheral lung lesions unreachable by conventional bronchoscopy in high-risk patients. J Bronchology Interv Pulmonol. 2011 Apr;18(2):133-7. doi: 10.1097/LBR.0b013e318216cee6. PMID 23169081
- [Background] Mukherjee S, Chacey M. Diagnostic Yield of Electromagnetic Navigation Bronchoscopy Using a Curved-tip Catheter to Aid in the Diagnosis of Pulmonary Lesions. J Bronchology Interv Pulmonol. 2017 Jan;24(1):35-39. doi: 10.1097/LBR.0000000000000326. PMID 27623421
- [Background] Lamprecht B, Porsch P, Wegleitner B, Strasser G, Kaiser B, Studnicka M. Electromagnetic navigation bronchoscopy (ENB): Increasing diagnostic yield. Respir Med. 2012 May;106(5):710-5. doi: 10.1016/j.rmed.2012.02.002. Epub 2012 Mar 3. PMID 22391437
- [Background] Rivera MP, Mehta AC, Wahidi MM. Establishing the diagnosis of lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e142S-e165S. doi: 10.1378/chest.12-2353. PMID 23649436